CLINICAL TRIAL: NCT04130230
Title: Safety and Efficacy of Neostigmine Infusion as Adjuvant Therapy in Sepsis and Septic Shock
Brief Title: Adjuvant Use of Neostigmine in Sepsis and Septic Shock.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mona Mohammed El-Tamalawy, Assistant lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-3
Record Dates: First submitted 2019-10-08; First posted 2019-10-17 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Sepsis, Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Neostigmine; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neostigmine group (Experimental): This arm will receive -in addition to standard therapy for sepsis and septic shock-Neostigmine methylsulfate ampoule diluted in normal saline, and administered as continuous infusion for five days. The rate of infusion is 0.2 mg/hr.
  Interventions: Drug: Neostigmine
- Standard group (Placebo Comparator): This arm will receive the standard therapy for sepsis and septic shock only and followed for five days.
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Neostigmine — Neostigmine continuous infusion plus standard therapy for sepsis and septic shock.
  Other Names: Choline esterase inhibitor
  Arms: Neostigmine group
Drug: Standard therapy — Standard therapy for sepsis and septic shock
  Arms: Standard group

SUMMARY:
The inflammatory response represents an important, central component of sepsis. Therefore, it is believed that blunting inflammation will decrease mortality. In vivo test series with mice that had undergone cecal ligation and puncture (recognized sepsis model), physostigmine salicylate significantly inhibited the release of various cytokines (tumor necrosis factor α, interleukin1β, and interleukin 6). These results were similar to those obtained by vagus nerve stimulation.

In animal sepsis model using physostigmine not only decreased inflammation but also, diminished the decrease in blood pressure following infection.

Animals treated with the peripheral choline esterase inhibitor neostigmine showed no difference compared with physostigmine-treated animals. Therefore, this study aims to investigate the efficacy of choline esterase inhibitors as adjuvant therapy in patients with sepsis or septic shock. Outcome measures include: percentage reduction in procalcitonin blood level, percentage of patients achieving significant reduction in procalcitonin levels, Mean Sequential Organ Failure Assessment score, percentage decrease in lactate dehydrogenase blood level, length of stay in hospital intensive care unit, and in hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years.
* Patients diagnosed with sepsis or septic shock according to Third International Consensus Definitions for Sepsis and Septic Shock mentioned above.
* Patients who have ≥ 2 of the following four criteria plus documented infection:

  1. Fever ≥ 38 °C or hypothermia ≤ 36 °C.
  2. Tachycardia ≥ 100/min.
  3. Tachypnea ≥ 20/min or hyperventilation.
  4. Leukocytosis ≥ 12000/mm3 or leukopenia ≤ 4000/mm3 or ≥ 10% immature neutrophils in the differential count.

Exclusion criteria:

* Known hypersensitivity to choline esterase inhibitors.
* Known absolute contra-indications against choline esterase inhibitors such as, myotonic dystrophy; depolarization block by depolarizing muscle relaxants; intoxication by irreversibly acting cholinesterase inhibitors; closed craniocerebral trauma; obstruction in the gastrointestinal tract (mechanical constipation); obstruction in the urinary tract (mechanical urinary retention)
* Known relative contraindications against choline esterase inhibitors: bronchial asthma; bradycardia; AV-conduction disturbances.
* Having undergone solid organ transplantation.
* Pregnant and lactating women.
* Participation in another clinical trial.
* Presence of primary or concomitant illness, impending death.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Sequential organ failure assessment (SOFA score) | Change from baseline SOFA score at five days
  Increase in SOFA score is associated with worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mamdouh M El-Shishtawy, Professor, Study Chair — Faculty of Pharmacy-Mansoura University
Locations (1):
- Tanta University Hospital, Tanta, EL-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Tamalawy MM, Soliman MM, Omara AF, Rashad A, Ibrahim OM, El-Shishtawy MM. Efficacy and Safety of Neostigmine Adjunctive Therapy in Patients With Sepsis or Septic Shock: A Randomized Controlled Trial. Front Pharmacol. 2022 Mar 7;13:855764. doi: 10.3389/fphar.2022.855764. eCollection 2022. PMID 35330830